CLINICAL TRIAL: NCT00002939
Title: A Phase I Trial of Dose Escalated Irinotecan (CPT-11) With Paclitaxel in Patients With Metastatic or Recurrent Malignancies
Brief Title: Irinotecan and Paclitaxel in Treating Patients With Metastatic or Recurrent Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8380; UCCRC-8380; NCI-G97-1166
Record Dates: First submitted 1999-11-01; First posted 2004-04-29 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Irinotecan; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel in combination with Irinotecan (Experimental): The first study cohort will receive 60 mg/m2 of paclitaxel on cycle days 1, 8, and 15 as a 1 hr infusion. Immediately following paclitaxel, 30 mg/m2 irinotecan will be administered as a 90 minute intravenous infusion. Irinotecan doses will be administered in an identical infusion schedule on days 8 and 15 of each treatment cycle.
  Interventions: Drug: irinotecan hydrochloride; Drug: paclitaxel

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of irinotecan and paclitaxel in treating patients with metastatic or recurrent cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) of irinotecan administered in combination with paclitaxel in patients with metastatic or recurrent malignancies. II. Evaluate the toxicity and safety of this combination regimen in this patient population. III. Determine the pharmacokinetic profile of irinotecan in combination with paclitaxel on a weekly schedule and if the sequence of administration influences irinotecan pharmacokinetics in these patients. IV. Determine pharmacodynamic models of irinotecan and its SN-38 and SN-38G metabolites when administered in this weekly combination schedule.

OUTLINE: This is a dose escalation study of irinotecan. Patients receive irinotecan IV concurrently with paclitaxel IV weekly. Patients demonstrating stable disease or partial or complete clinical response continue with treatment as long as dose limiting toxicities are not observed and adequate performance status is maintained. Cohorts of 3 patients receive escalating doses of irinotecan until the maximum tolerated dose is determined or 150 mg/m2 is reached.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed non hematologic malignancy refractory to standard therapy, or for which no known effective therapies exist

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 3 months Hematopoietic: Platelet count at least 100,000/mm3 Absolute neutrophil count at least 2,000/mm3 Absolute lymphocyte count at least 1,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminase no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 1.4 mg/dL Cardiovascular: No myocardial infarction within 6 months No current, uncontrolled cardiac arrhythmias Other: No history of anaphylactic reactions Not pregnant Fertile patients must use effective contraception No serious uncontrolled, concurrent medical disorder

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior paclitaxel allowed No prior irinotecan At least 4 weeks since prior chemotherapy Endocrine therapy: No concurrent steroids Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 1996-11; Primary Completion 2001-02 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose | 3 weeks
  Determine the maximum tolerated dose of irinotecan administered on a weekly schedule with fixed-dose weekly paclitaxel.

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L. Kindler, MD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States